CLINICAL TRIAL: NCT02801578
Title: A Pilot Study of Different Doses of Ibrutinib in Participants With Chronic Lymphocytic Leukemia (CLL)
Brief Title: A Study of Different Doses of Ibrutinib in Participants With Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0226; NCI-2016-01091 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-05-27; First posted 2016-06-16 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Malignant neoplasms stated as primary lymphoid haematopoietic; Ibrutinib; PCI-32765; Imbruvica; Pharmacodynamics
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib (Experimental): Participants take Ibrutinib capsules by mouth every day for 3, 28 day cycles.
  During Cycle 1, participants receive the highest dose of Ibrutinib by taking 3 capsules each day. During Cycle 2, participants receive the second-highest dose and will take 2 capsules each day. During Cycle 3, participant takes the lowest dose of Ibrutinib and takes 1 capsule each day.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Cycle 1 daily dose of ibrutinib is 420 mg (3 capsules), in the second cycle 280 mg (2 capsules), and in the third cycle 140 mg (1 capsule).
  Other Names: PCI-32765; Imbruvica

SUMMARY:
Ibrutinib is currently FDA approved and commercially available for the treatment of CLL. However, some researchers think the approved dose may be unnecessarily high.

The goal of this clinical research study is to compare 3 different daily doses of ibrutinib to learn how these doses affect the disease and your body. Researchers think that if a lower dose of ibrutinib can be found to be as effective as the currently approved dose this may help to lower the risk of side effects.

DETAILED DESCRIPTION:
Study Drug Administration:

Each study cycle is 28 days.

If you are found to be eligible to take part in this study, you will take ibrutinib capsules by mouth every day for 3 cycles. Each dose of ibrutinib should be taken at about the same time, either with or without food.

During Cycle 1, you will receive the highest dose of ibrutinib (the dose that is currently FDA approved). You will take 3 capsules each day during Cycle 1. During Cycle 2, you will receive the second-highest dose and you will take 2 capsules each day. During Cycle 3, you will take the lowest dose of ibrutinib and you will take 1 capsule each day.

You must swallow the ibrutinib capsules whole without opening, breaking, or chewing them.

You will be given a study drug diary to keep track of each dose of ibrutinib taken, including the time the dose was taken, any missed or vomited doses and the reason for missing the dose, and any doses that you vomited.

Study Visits:

On Days 1, 8 and 28 of each cycle blood (about 1-2 tablespoons total) will be drawn before your dose of ibrutinib and then at 4 and 24 hours after your dose for pharmacodynamic (PD) and pharmacokinetic (PK) testing, to help researchers understand how ibrutinib works in the body, and to learn if the dose you are taking is as effective as other doses (Exception: there will be no 4-hour blood draw on day 28). PK testing measures the amount of study drug in the body at different time points. PD testing measures how the level of study drug in your body may affect the disease. You will need to return to the clinic on the following day (Days 2, 9 and 29 of each cycle [Day 1 of the next cycle]) for the last blood draw.

On Day 28 of each cycle:

* You will have a physical exam
* Blood (about 1-2 tablespoons) will be drawn for routine tests.
* You will have an EKG.

Length of Study:

You may receive ibrutinib on this study for up to 3 cycles. After this time, you will continue treatment for CLL as directed by your doctor. This may or may not include ibrutinib. If you do continue to take ibrutinib after the study is over, your doctor will determine the best dose for you to be taking.

You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation in this study will be over after your last dose of ibrutinib (after the end of Cycle 3).

This is an investigational study. Ibrutinib is FDA approved and commercially available for the treatment of CLL. It is considered investigational to compare 3 different doses of ibrutinib. The study doctor can explain how the study drug is designed to work.

Up to 12 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of CLL (any stage) with ALC >/= 20 x 109/l, requiring therapy.
2. Able to receive ibrutinib through commercial supply, i.e., insured patients meeting FDA-approved indications.
3. Age >/=18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Adequate end organ function, defined as the following: total bilirubin </= 1.5 x upper limit of normal (ULN, unless due to Gilbert syndrome, in which case it should be </= 3.0 x ULN), ALT and AST </= 2.5 x ULN, CrCL >/= 25 ml/min.
6. Able to understand and sign the IRB-approved informed consent document for this trial.
7. Women of childbearing potential (WOCBP) must practice 2 effective methods of birth control during the course of the study. Male patients who are partners of WOCBP should also practice an effective method of contraception. Effective methods of birth control include diaphragm or condoms with spermicidal foam or jelly, birth control pills (BCPs), injections or patches, intra-uterine devices (IUDs) and surgical sterilization. Postmenopausal women must be amenorrheic for >/= 12 months to be considered of non-childbearing potential, Women and men must continue birth control for the duration of the trial and >/= 3 months after the last dose of study drug, All WOCBP MUST have a negative pregnancy test prior to beginning ibrutinib on study.
8. Patients should have discontinued any and all other therapy for CLL >/= 48 hours prior to start of study therapy and recovered from any toxicity due to these therapies to grade </= 1.

Exclusion Criteria:

1. Previous treatment with ibrutinib.
2. Current therapy with warfarin or other anticoagulants at therapeutic doses, e.g., low molecular weight heparin, fondaparinux, dabigatran, rivaroxaban, apixaban or edoxaban that are unable to be discontinued.
3. Active gastrointestinal conditions that are expected to impair absorption of orally administered medications.
4. Active, uncontrolled infection.
5. History of hypersensitivity to ibrutinib.
6. Pregnancy or lactation.
7. Patients with leukemic involvement of the central nervous system.
8. Patients who currently have or have a history of the following within 6 months preceding study entry are not eligible: Unstable angina (UA) or myocardial infarction (MI), Clinically significant atrial or ventricular arrhythmias (e.g., AF, atrial flutter, ventricular tachycardia, ventricular fibrillation, or torsades de pointes), New York Heart Association (NYHA) class III or IV heart failure.
9. Patients on strong CYP3A inducers or inhibitors that are unable to be discontinued. The list of drugs that interact with cytochrome P450 enzymes can be found online at: http://medicine.iupui.edu/clinpharm/DDIs/ClinicalTable.aspx

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prithviraj Bose, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chen LS, Bose P, Cruz ND, Jiang Y, Wu Q, Thompson PA, Feng S, Kroll MH, Qiao W, Huang X, Jain N, Wierda WG, Keating MJ, Gandhi V. A pilot study of lower doses of ibrutinib in patients with chronic lymphocytic leukemia. Blood. 2018 Nov 22;132(21):2249-2259. doi: 10.1182/blood-2018-06-860593. Epub 2018 Sep 25. PMID 30254130
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 2016 to June 2017
Groups:
- Ibrutinib: Participants take Ibrutinib capsules by mouth every day for 3, 28 day cycles.
  During Cycle 1, participants receive the highest dose of Ibrutinib by taking 3 capsules each day. During Cycle 2, participants receive the second-highest dose and will take 2 capsules each day. During Cycle 3, participant takes the lowest dose of Ibrutinib and takes 1 capsule each day.
  Ibrutinib: Cycle 1 daily dose of ibrutinib is 420 mg (3 capsules), in the second cycle 280 mg (2 capsules), and in the third cycle 140 mg (1 capsule).
Period: Overall Study
Arm/Group | Ibrutinib
Started | 11
Completed | 9
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 68 [52 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Participants With >/= 95 % Bruton's Tyrosine Kinase (BTK) Occupancy
Description: BTK occupancy level measured by fluorescent affinity probe just before dosing and at 4 and 24 hours post-dosing on days 1, 8, and 28 (but before the first dose of the next cycle) of each cycle.
Time Frame: 3 cycles, up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib
Number analyzed (Participants) | 9
Participants | 8

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Ibrutinib
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib (N=11)
Surgical Procedure (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib (N=11)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT02801578/Prot_SAP_000.pdf